CLINICAL TRIAL: NCT02412098
Title: A Phase 1, Open-Label, Parallel-Group, Adaptive, Single Dose Study to Evaluate the Pharmacokinetics of GS-6615 in Subjects With Normal and Impaired Hepatic Function
Brief Title: Pharmacokinetics of Eleclazine in Adults With Normal and Impaired Hepatic Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-372-1048; 2014-005266-30 (EudraCT Number)
Record Dates: First submitted 2015-03-11; First posted 2015-04-08 (Estimated); Results first posted 2019-07-29 (Actual); Last update posted 2019-07-29 (Actual); Status verified 2019-05

CONDITIONS: Long QT Syndrome
Keywords: Hepatic Impairment
MeSH Terms: conditions — Long QT Syndrome | interventions — eleclazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Moderate Hepatic Impairment (Cohort 1) (Experimental): Participants with moderate hepatic impairment and matched healthy controls will receive a single dose of eleclazine 30 mg (5 x 6 mg tablets).
  Interventions: Drug: Eleclazine
- Severe Hepatic Impairment (Cohort 2) (Experimental): Participants with severe hepatic impairment and matched healthy controls will receive a single dose of eleclazine 30 mg (5 x 6 mg tablets).
  Interventions: Drug: Eleclazine
- Mild Hepatic Impairment (Cohort 3) (Experimental): Participants with mild hepatic impairment and matched healthy controls will receive a single dose of eleclazine 30 mg (5 x 6 mg tablets).
  Interventions: Drug: Eleclazine

INTERVENTIONS:
Drug: Eleclazine — Eleclazine tablets administered orally
  Other Names: GS-6615

SUMMARY:
The primary objective of this study is to evaluate the pharmacokinetic (PK) profile of oral eleclazine and its metabolite, GS-623134, in participants with normal and impaired hepatic function. Participants in the healthy control group will be matched to participants with impaired hepatic function by age (± 5 years), gender, and body mass index (± 10%).

ELIGIBILITY:
Inclusion Criteria:

All participants:

* Be a nonsmoker or consume < 20 cigarettes per day
* Have a calculated body mass index (BMI) from 18 to 36 kg/m^2, inclusive, at study screening
* Have a creatinine clearance (CrCl) ≥ 60 mL/min (using the Cockcroft-Gault method) based on serum creatinine and actual body weight as measured at screening
* Have either a normal 12-lead electrocardiogram (ECG) or one with abnormalities that are considered clinically insignificant by the investigator
* Screening labs within defined thresholds

Participants with mild, moderate, or severe hepatic impairment must also meet the following additional inclusion criteria:

* Must have diagnosis of chronic (> 6 months), stable hepatic impairment with no clinically significant changes within 3 months (90 days) prior to study drug administration (Day 1)
* Individuals with severe hepatic impairment must have a score on the Child-Pugh-Turcotte scale of 10-15 at screening. If an individual's score changes during the course of the study, the score at screening will be used for classification.
* Individuals with moderate hepatic impairment must have a score on the Child-Pugh-Turcotte scale of 7-9 at screening. If an individual's score changes during the course of the study, the score at Screening will be used for classification.
* Individuals with mild hepatic impairment must have a score on the Child-Pugh-Turcotte scale of 5-6 at screening. If an individual's score changes during the course of the study, the score at screening will be used for classification.

Exclusion Criteria:

* Pregnant or lactating females
* History of meningitis or encephalitis, epilepsy, seizures, migraines, tremors, myoclonic jerks, narcolepsy, obstructive sleep apnea, anxiety, syncope, head injuries or a family history of seizures
* Presence or history of cardiovascular disease (including history of myocardial infarction based on ECG and/or clinical history, any history of ventricular tachycardia, congestive heart failure, cardiomyopathy, or left ventricular ejection fraction < 40%), cardiac conduction abnormalities, a family history of Long QT Syndrome, or unexplained death in an otherwise healthy individual between the ages of 1 and 30 years
* Syncope, palpitations, or unexplained dizziness
* Implanted defibrillator or pacemaker
* Are unable to comply with study requirements or are otherwise believed, by the study investigator, to be inappropriate for study participation for any reason

Participants with mild, moderate, or severe hepatic impairment must also meet the following additional exclusion criteria:

* Active hepatitis B virus (HBV) infection. Individuals who have HBsAg are ineligible
* Requires paracentesis > 1 time per month
* Severe (grade 3 or 4) encephalopathy as judged by the investigator
* History of gastric or esophageal variceal bleeding within the past 6 months and for which varices have not been adequately treated with medication and/or surgical procedures

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2015-03-19 (Actual); Primary Completion 2016-04-22 (Actual); Study Completion 2016-04-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (7):
- United States (4):
  - Miami, Florida
  - Orlando, Florida
  - Minneapolis, Minnesota
  - Kansas City, Missouri
- München, Germany
- Auckland, New Zealand
- Bucharest, Romania

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in United States, Romania, Germany, and New Zealand. The first participant was screened on 19 March 2015. The last study visit occurred on 22 April 2016.
Pre-assignment Details: 91 participants were screened. No participants were enrolled in the severe hepatic impairment (cohort 2) arm.
Groups:
- Moderate Hepatic Impairment (Cohort 1): Participants with moderate hepatic impairment received a single dose of eleclazine 30 mg (5 x 6 mg tablets) on Day 1.
- Mild Hepatic Impairment (Cohort 3): Participants with mild hepatic impairment received a single dose of eleclazine 30 mg (5 x 6 mg tablets) on Day 1.
- Normal Hepatic Function: Participants with normal hepatic function received a single dose of eleclazine 30 mg (5 x 6 mg tablets) on Day 1.
Period: Overall Study
Arm/Group | Moderate Hepatic Impairment (Cohort 1) | Mild Hepatic Impairment (Cohort 3) | Normal Hepatic Function
Started | 14 | 14 | 21
Completed | 14 | 14 | 21
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set included all enrolled participants who received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Moderate Hepatic Impairment (Cohort 1) | Mild Hepatic Impairment (Cohort 3) | Normal Hepatic Function | Total
Number analyzed (Participants) | 14 | 14 | 21 | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (5.3) | 57 (8.9) | 55 (6.9) | 56 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 7 | 15
  Male | 10 | 10 | 14 | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 1 | 9 | 15
  Not Hispanic or Latino | 9 | 13 | 12 | 34
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 3 | 6
  White | 12 | 12 | 18 | 42
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13 | 6 | 16 | 35
  Romania | 0 | 4 | 2 | 6
  Germany | 0 | 2 | 2 | 4
  New Zealand | 1 | 2 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: PK (Pharmacokinetic) Parameter: AUCinf of Eleclazine
Description: AUCinf was defined as the concentration of drug extrapolated to infinite time (area under the plasma concentration versus time curve extrapolated to infinite time).
Time Frame: Predose and 0.5, 1, 2, 3, 4, 6, 8, 10, 14, 24, 36, 48, 72, 96, 120 hours on Day 1 and approximately the same time in the morning as predose of Day 1 on Days 15, 29, 43, and 57
Population: PK Analysis Set included all enrolled participants who received at least one dose of eleclazine and had at least one evaluable PK concentration value reported by the PK laboratory for the corresponding analyte. Healthy control participants may participate in more than one cohorts.
Measure: Geometric Mean (95% Confidence Interval); unit: h*ng/mL
Groups:
- Normal Hepatic Function (Matched Control for Cohort 1): Normal hepatic function (matched control for Cohort 1) included participants that served as controls for participants with moderate hepatic impairment.
- Normal Hepatic Function (Matched Control for Cohort 3): Normal hepatic function (matched control for Cohort 3) included participants that served as controls for participants with mild hepatic impairment.
Arm/Group | Moderate Hepatic Impairment (Cohort 1) | Mild Hepatic Impairment (Cohort 3) | Normal Hepatic Function (Matched Control for Cohort 1) | Normal Hepatic Function (Matched Control for Cohort 3)
Number analyzed (Participants) | 14 | 14 | 14 | 14
h*ng/mL | 42503.2 [23983.8 to 75322.7] | 50064.7 [31758.4 to 78923.2] | 57795.9 [37994.2 to 87917.5] | 39173.2 [23050.5 to 66573.2]
Statistical Analysis 1: Comparison: Moderate Hepatic Impairment (Cohort 1) vs Normal Hepatic Function (Matched Control for Cohort 1); An analysis of variance (ANOVA) appropriate for a parallel design was fit to the natural logarithmic transformation of eleclazine AUCinf; Test type: Other; Geometric Least Square Mean (GLSM) Ratio = 73.54, 90% CI 2-sided [41.92 to 129.01] — A 90% CI was constructed for the GLSM ratio of AUCinf in the hepatic impairment group versus matched control
Statistical Analysis 2: Comparison: Mild Hepatic Impairment (Cohort 3) vs Normal Hepatic Function (Matched Control for Cohort 3); [analysis description as in outcome 1, analysis 1]; Test type: Other; GLSM Ratio (%) = 127.80, 90% CI 2-sided [73.57 to 222.01] — A 90% CI was constructed for the GLSM ratio of AUCinf in the hepatic impairment group versus matched control

2. Primary Outcome: PK Parameter: AUCinf of GS-623134 (Metabolite of Eleclazine)
Description: as for outcome 1
Time Frame: as for outcome 1
Population: Participants in the PK Analysis Set with available data were analyzed. Healthy control participants may participate in more than one cohorts.
Measure: Geometric Mean (95% Confidence Interval); unit: h*ng/mL
Arm/Group | Moderate Hepatic Impairment (Cohort 1) | Mild Hepatic Impairment (Cohort 3) | Normal Hepatic Function (Matched Control for Cohort 1) | Normal Hepatic Function (Matched Control for Cohort 3)
Number analyzed (Participants) | 7 | 10 | 8 | 12
h*ng/mL | 1880.0 [980.5 to 3604.4] | 1983.2 [1238.3 to 3176.0] | 2326.2 [1497.0 to 3614.9] | 2697.4 [2023.1 to 3596.5]
Statistical Analysis 1: Comparison: Moderate Hepatic Impairment (Cohort 1) vs Normal Hepatic Function (Matched Control for Cohort 1); ANOVA appropriate for a parallel design was fit to the natural logarithmic transformation of GS-623134 AUCinf; Test type: Other; GLSM Ratio (%) = 80.82, 90% CI 2-sided [45.11 to 144.79] — A 90% CI was constructed for the GLSM ratio of AUCinf in the hepatic impairment group versus matched control
Statistical Analysis 2: Comparison: Mild Hepatic Impairment (Cohort 3) vs Normal Hepatic Function (Matched Control for Cohort 3); Test type: Other; ANOVA appropriate for a parallel design was fit to the natural logarithmic transformation of GS-623134 AUCinf; GLSM Ratio (%) = 73.52, 90% CI 2-sided [47.83 to 113.02] — A 90% CI was constructed for the GLSM ratio of AUCinf in the hepatic impairment group versus matched control

3. Primary Outcome: PK Parameter: Cmax of Eleclazine
Description: Cmax was defined as the maximum observed concentration of drug in plasma.
Time Frame: as for outcome 1
Population: Participants in the PK Analysis Set were analyzed. Healthy control participants may participate in more than one cohorts.
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Moderate Hepatic Impairment (Cohort 1) | Mild Hepatic Impairment (Cohort 3) | Normal Hepatic Function (Matched Control for Cohort 1) | Normal Hepatic Function (Matched Control for Cohort 3)
Number analyzed (Participants) | 14 | 14 | 14 | 14
ng/mL | 214.9 [169.4 to 272.5] | 338.1 [283.6 to 403.1] | 322.9 [279.4 to 373.1] | 331.3 [273.1 to 401.9]
Statistical Analysis 1: Comparison: Moderate Hepatic Impairment (Cohort 1) vs Normal Hepatic Function (Matched Control for Cohort 1); ANOVA appropriate for a parallel design was fit to the natural logarithmic transformation of eleclazine Cmax; Test type: Other; GLSM Ratio (%) = 66.55, 90% CI 2-sided [53.33 to 83.04] — A 90% CI was constructed for the GLSM ratio of Cmax in the hepatic impairment group versus matched control
Statistical Analysis 2: Comparison: Mild Hepatic Impairment (Cohort 3) vs Normal Hepatic Function (Matched Control for Cohort 3); ANOVA appropriate for a parallel design was fit to the natural logarithmic transformation of eleclazine Cmax; Test type: Other; GLSM Ratio (%) = 102.06, 90% CI 2-sided [83.03 to 125.45] — A 90% CI was constructed for the GLSM ratio of Cmax in the hepatic impairment group versus matched control

4. Primary Outcome: PK Parameter: Cmax of GS-623134 (Metabolite of Eleclazine)
Description: Cmax was defined as the maximum observed concentration of drug in plasma.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Moderate Hepatic Impairment (Cohort 1) | Mild Hepatic Impairment (Cohort 3) | Normal Hepatic Function (Matched Control for Cohort 1) | Normal Hepatic Function (Matched Control for Cohort 3)
Number analyzed (Participants) | 11 | 13 | 14 | 14
ng/mL | 4.9 [3.2 to 7.7] | 7.3 [4.6 to 11.4] | 6.5 [5.0 to 8.4] | 10.2 [7.0 to 15.0]
Statistical Analysis 1: Comparison: Moderate Hepatic Impairment (Cohort 1) vs Normal Hepatic Function (Matched Control for Cohort 1); ANOVA appropriate for a parallel design was fit to the natural logarithmic transformation of GS-623134 Cmax; Test type: Other; GLSM Ratio (%) = 76.24, 90% CI 2-sided [50.65 to 114.77] — A 90% CI was constructed for the GLSM ratio of Cmax in the hepatic impairment group versus matched control
Statistical Analysis 2: Comparison: Mild Hepatic Impairment (Cohort 3) vs Normal Hepatic Function (Matched Control for Cohort 3); ANOVA appropriate for a parallel design was fit to the natural logarithmic transformation of GS-623134 Cmax; Test type: Other; GLSM Ratio (%) = 71.06, 90% CI 2-sided [44.59 to 113.25] — A 90% CI was constructed for the GLSM ratio of Cmax in the hepatic impairment group versus matched control

5. Secondary Outcome: Number of Participants Experiencing Treatment-Emergent Adverse Events
Description: Treatment-emergent adverse events (AEs) are defined as one or both of the following:
  * Any AEs with an onset date on or after the study drug start date and no later than 30 days after permanent discontinuation of study drug.
  * Any AEs leading to premature discontinuation of study drug.
Time Frame: First dose date up to 31 days
Population: Safety Analysis Set included all enrolled participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Moderate Hepatic Impairment: Participants with moderate hepatic impairment received a single dose of eleclazine 30 mg (5 x 6 mg tablets) on Day 1.
- Mild Hepatic Impairment: Participants with mild hepatic impairment received a single dose of eleclazine 30 mg (5 x 6 mg tablets) on Day 1.
Arm/Group | Moderate Hepatic Impairment | Mild Hepatic Impairment | Normal Hepatic Function
Number analyzed (Participants) | 14 | 14 | 21
Participants | 6 | 8 | 3

6. Secondary Outcome: Number of Participants Experiencing Clinical Laboratory Abnormalities
Description: Treatment-emergent laboratory abnormalities reported as an adverse event (AE) or serious adverse event (SAE) are presented. Laboratory abnormalities that required medical or surgical intervention or led to study drug interruption, modification, or discontinuation were recorded as an AE or SAE, as applicable, and are reported here. Laboratory abnormalities without clinical significance were not recorded as AEs or SAEs and therefore, are not being reported.
Time Frame: First dose date up to 31 days
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Moderate Hepatic Impairment | Mild Hepatic Impairment | Normal Hepatic Function
Number analyzed (Participants) | 14 | 14 | 21
Participants
  Blood Creatinine Increased | 0 | 1 | 0
  Gamma-glutamyltransferase Increased | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: First dose date up to 31 days
Description: Safety Analysis Set included all enrolled participants who received at least one dose of study drug.
Arm/Group | Moderate Hepatic Impairment | Mild Hepatic Impairment | Normal Hepatic Function
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14 | 0/21
Other Adverse Events (participants affected / at risk) | 6/14 | 8/14 | 3/21
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Moderate Hepatic Impairment (N=14) | Mild Hepatic Impairment (N=14) | Normal Hepatic Function (N=21)
Atrial flutter (Cardiac disorders) | 0 | 1 | 0
Atrioventricular block first degree (Cardiac disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 0
Electrocardiogram PR prolongation (Investigations) | 0 | 1 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 1
Headache (Nervous system disorders) | 1 | 0 | 0
Somnolence (Nervous system disorders) | 3 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 2 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years